CLINICAL TRIAL: NCT06009601
Title: Are Pectus Deformities a Projection of Spinal Pathologies?The Relationship Between Pectus Deformities and Spinal Pathologies
Brief Title: The Relationship Between Pectus Deformities and Spinal Pathologies
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 397
Record Dates: First submitted 2023-01-11; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-06

CONDITIONS: Pectus Deformity of Chest; Spinal Deformity
Keywords: Pectus Excavatum; Pectus Carinatum; Scoliosis; Kyphosis; Lordosis
MeSH Terms: conditions — Funnel Chest; Pectus Carinatum; Scoliosis; Kyphosis; Lordosis | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged 3-18 years who were diagnosed with pectus deformity: Pectus study forms consisting of clinical and radiological measurements of patients aged 3-18 years who applied to the outpatient clinic with chest deformity will be filled in in detail.
  Interventions: Diagnostic Test: Pectus Study Form; Diagnostic Test: Adams Test; Diagnostic Test: Scoliosis Graphy; Diagnostic Test: Pulmonary function test

INTERVENTIONS:
Diagnostic Test: Pectus Study Form — Pectus study forms consisting of clinical and radiological measurements of patients aged 3-18 years who applied to the outpatient clinic with chest deformity will be filled in in detail.
  In addition, this study form includes 'Quality of Life Evaluation Form in Pectus Deformity', 'Social Comparison Scale', 'Sleep Disorder Scale for Children', 'Anxiety Disorders Screening Scale in Children', 'Pediatric Quality of Life Questionnaire' designed for patients and their relatives. PedsQL)', 'SRS-22 Patient Questionnaire', 'Beck Anxiety Scale' and 'Informed Consent Form' designed for patients and their relatives.
Diagnostic Test: Adams Test — Adams test (forward bending test) (+) was measured by Bunnell scoliometer (scoliosis assessment tool) and ATR (angle of trunk rotation angle) values were 7 degrees in patients who meet the inclusion criteria will be included in the study by filling out an informed consent form
  Other Names: Forward Bending Test
Diagnostic Test: Scoliosis Graphy — ATR (angle of trunk rotation) values above 7 degrees on bunnell scoliometer were determined. Afterwards, patients who meet the inclusion criteria will be included in the study by filling out an informed consent form and a scoliosis graphy will be requested.
  Coronal, sagittal balance; coronal and sagittal cobb angles will be measured from posterior-anterior (PA) (posterior-anterior) and lateral (lateral) scoliosis radiographs.
  Other Names: Orthoroentgenogram
Diagnostic Test: Pulmonary function test — Pulmonary function tests (PFTs) are noninvasive tests that show how well the lungs are working. The tests measure lung volume, capacity, rates of flow, and gas exchange. This information can help your healthcare provider diagnose and decide the treatment of certain lung disorders.
  There are 2 types of disorders that cause problems with air moving in and out of the lungs:
  Obstructive. This is when air has trouble flowing out of the lungs due to airway resistance. This causes a decreased flow of air.
  Restrictive. This is when the lung tissue and/or chest muscles can't expand enough. This creates problems with air flow, mostly due to lower lung volumes.
  Other Names: Spirometry Function Test

SUMMARY:
Pectus deformities are common anterior chest wall pathologies. Pectus excavatum is the most common chest deformity with an incidence of 0.1-0.3%. Although the incidence of adolescent idiopathic scoliosis (AIS) is 0.2-3% in the community, some studies show that this rate rises to 17.61-25.58% when it is associated with pectus deformity. While the pectus excavatum rotates the heart to the left with its ribs and cartilages, it pushes the thoracic vertebra to the right side with the internal counterforce created by the heart, which has been shown to push the spine to the right with an asymmetric horizontal force in scoliosis patients with pectus deformity.

Based on this, in study, investigators aimed to determine whether there is any relationship between pectus deformities and spinal pathologies, and if there is a relationship, with which pathology it is most common, whether the type of scoliosis seen in pectus deformities with a prominent scoliosis prevalence is a pectus-specific curve, and whether this curve seen in scoliosis is associated with pectus. To determine whether there is a footprint or not.

DETAILED DESCRIPTION:
The study was planned as a prospective cross-sectional study. Pectus study forms consisting of clinical and radiological measurements of the patients aged 3-18 years who applied to the outpatient clinic with chest deformity will be filled in in detail, and the Adams test (forward bending test) (+) will be measured by Bunnell scoliometer (scoliosis assessment tool) and ATR (angle of trunk rotation- trunk rotation) measurements. If ATR measurement is above 7 degrees on Bunnell scoliometer, patients who meet the inclusion criteria will be included in the study by filling in the informed consent form and a scoliosis radiograph will be requested (Independent of investigators' study, it is necessary to withdraw it in line with the 2016 recommendations of the International Scientific Society for Scoliosis Orthopedic and Rehabilitation Treatment (SOSORT).)

Coronal, sagittal balance, coronal and sagittal cobb angles will be measured from the scoliosis radiograph taken from the Posterior-Anterior (PA) (posterior-anterior) and lateral (side) films. Their relationship with chest deformities will be evaluated. All measurements will be made and recorded by two independent investigators As a result of the analysis, when the power is targeted as 95% and the error amount as 0.05, the minimum sample size required for investigators to find a significant difference between the means was determined as 36. Investigators formed a sample group of 40 people for our study, together with the fact that groups of 36 people were sufficient in terms of providing 95% power. Kappa statistical analysis will be used to determine intraobserver and interobserver variations.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with pectus deformity
* Be between 3-18 years old

Exclusion Criteria:

* Adult type scoliosis
* Congenital scoliosis
* Neuromuscular scoliosis
* Syndromic scoliosis
* Infantile idiopathic scoliosis
* Having surgery to the chest wall or spine
* People with connective tissue disease will not be included in the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pectus study forms consisting of clinical and radiological measurements of patients aged 3-18 years who applied to the outpatient clinic with chest deformity will be filled in in detail. Adams test (forward bending test) (+) was measured by Bunnell scoliometer (scoliosis assessment tool) and ATR (angle of trunk rotation angle) values were 5 degrees in those with BMI (Body Mass Index) above 85%. If it is below 85% and above 7 degrees, patients who meet the inclusion criteria will be included in the study by filling out an informed consent form and a scoliosis film will be requested. Scoliosis X-ray (orthorontgenogram) will be requested. Coronal, sagittal balance, coronal and sagittal cobb angles will be measured. Their relationship with chest deformities will be evaluated. All measurements will be made and recorded by two independent researchers.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-04-09 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Pectus Study Form | Within 1 week of applying to the scoliosis outpatient clinic
  In the Pectus Study Form, the clinical and radiological data of the patient will be evaluated. Coronal, sagittal balance and coronal and sagittal cobb angles of the patient will be measured in the scoliosis X-ray.
Pulmonary Function Test (PFT) | Within 1 week of applying to the scoliosis outpatient clinic
  Pulmonary function test measurements will be made for people with pectus deformity.Pulmonary function tests, or PFTs, measure how well the lungs work. For some of the test measurements, the client can breathe normally and quietly. Other tests require forced inhalation or exhalation after a deep breath. Sometimes, they will be asked to inhale a different gas or a medicine to see how it changes test results.
Body Aesthetic Clinical Evaluation (TRACE) | Within 1 week of applying to the scoliosis outpatient clinic
  Body Aesthetic Clinical Evaluation (TRACE) measurement will be performed.TRACE is a 12-point scale based on four sub-scales, shoulders (0-3), scapulae (0-2), hemi-thorax (0-2) and waist (0-4)

SECONDARY OUTCOMES:
Quality of Life Evaluation Form in Pectus Deformity | Within 1 week of applying to the scoliosis outpatient clinic
  This questionnaire, a self-assessment one, will assist clinicians who wish to assess body image and quality of life of patients with Pectus deformity. The PEEQ is a questionnaire used to assess the disease-speciﬁc quality of life of patients with PE and their parents. The questionnaire contains 12 items and the parent form contains 13 items. Each item receives a score between 1 and 4, with higher scores indicating a better quality of life. The questionnaire has subscales that indicate psychosocial and physical quality of life for both children and parents. The questions from 1 to 9 in the child form ask about psycho-social quality of life, while the questions 10-12 ask about physical quality of life. In the parents form, the questions from 1 to 8 ask about psychosocial quality of life, while the questions from 9 to13 ask about physical quality of life.
Social Comparison Scale | Within 1 week of applying to the scoliosis outpatient clinic
  This scale was developed by Allan and Gilbert (1995) to measure self-perceptions of social rank and relative social standing. This scale uses a semantic differential methodology and consists of 11 bipolar constructs. Participants are required to make a global comparison of themselves in relation to other people and to rate themselves along a ten-point scale. For example' the scale asks:
  In relationship to others I feel: Incompetent ->1 2 3 4 5 6 7 8 9 10 <- More competent The 11-items cover judgments concerned with rank' attractiveness and how well the person thinks they 'fit in' with others in society. Low scores point to feelings of inferiority and general low rank self-perceptions.
Sleep Disorder Scale for Children | Within 1 week of applying to the scoliosis outpatient clinic
  Sleep Disorder Scale for Children (SDSC) was designed both to evaluate specific sleep disorders in children, and to provide an overall measure of sleep disturbance suitable for use in clinical screening and research. Using factor analysis, developers Bruni and colleagues divided items into six categories representing some of the most common sleep diffi culties affecting adolescents and children: disorders of initiating and maintaining sleep, sleep breathing disorders, disorders of arousal/nightmares, sleep-wake transition disorders, disorders of excessive somnolence, and sleep hyperhidrosis (nighttime sweating).
Anxiety Disorders Screening Scale in Children | Within 1 week of applying to the scoliosis outpatient clinic
  Anxiety Disorders Screening Scale in Children (SCARED) is a child self-report instrument used to screen for childhood anxiety disorders including general anxiety disorder, separation anxiety disorder, panic disorder and social phobia. The SCARED consists of 41 items and 5 factors that parallel the DSM-IV classification of anxiety disorders.The Screen for Child Anxiety Related Emotional Disorders (SCARED) assesses a range of DSM-IV based anxiety symptomatology. More specifically, it taps symptoms of panic disorder (13 items), generalised anxiety disorder (9 items), social phobia (9 items), separation anxiety disorder (12 items), obsessive-compulsive disorder (9 items), post-traumatic stress disorder (4 items), and specific phobia (15 items). The SCARED-71 consists of 71 items rated on a three-point scale (0 = almost never, 1 = sometimes, 2 = often). The minimum score that could be obtained is 0 and the maximum score that could be obtained is 142.
The Pediatric Quality of Life Inventory | Within 1 week of applying to the scoliosis outpatient clinic
  The Pediatric Quality of Life Inventory (PedsQL) is a 23-item generic health status instrument with parent and child forms that assesses five domains of health (physical functioning, emotional functioning, psychosocial functioning, social functioning, and school functioning) in children and adolescents ages 2 to 18. Each item of the instrument is scored on a 5-point scale from 0- 4 for ages 8-18, (0 = never a problem, 1 = almost never a problem, 2 = sometimes a problem, 3 = often a problem, 4 = almost always a problem) ad 3-point scale for young child self reporting (ages 5- 7) as following (0 = not at all a problem, 2 = sometimes a problem, 4 = a lot of a problem) the large score means worst symptoms , scores are linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0) in which high score means better condition
Scoliosis Research Society Score | Within 1 week of applying to the scoliosis outpatient clinic
  The SRS-22r is a validated questionnaire intended to assess outcomes in patients with idiopathic scoliosis after spinal surgery. The first version, developed by the Scoliosis Research Society in 1999, had 24 items, and this was reduced to 22 items (accompanied by a name change) in the course of 3 major updates.The SRS-22 contains 22 questions covering 5 domains: function/activity 5 items; pain 5 items; self-perceived image 5 items; mental health 5 items; and satisfaction with treatment 2 items. Each item is scored from 1 (worst) to 5 (best). Each domain has a total sum score ranging from 5 to 25, except for satisfaction, which ranges from 2 to 10. The sum of the first 4 domains gives a maximum subtotal of 100, and when the satisfaction domain is included, the maximum total is 110
Beck Anxiety Scale | Within 1 week of applying to the scoliosis outpatient clinic
  The Beck Anxiety Inventory (BAI), created by Aaron T. Beck and other colleagues, is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in adolescents and adults ages 17 and older.The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. The standardized cutoffs are:0-7: Minimal, 8-15: Mild, 16-25: Moderate,and 26-63: Severe

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Guneser Gulec, MD, Study Chair — Gaziosmanpasa Training and Research Hospital Physical Rehabilitation Department; Ebru Yilmaz Yalcinkaya, Prof, Study Director — Gaziosmanpasa Training and Research Hospital Physical Rehabilitation Department
Locations (1):
- Deniz, Gaziosmanpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study will be available on request from the corresponding author (EG). The data will not be publicly available due to their containing information that could compromise the privacy of research participants.

REFERENCES:
- [Result] Zhong W, Ye J, Feng J, Geng L, Lu G, Liu J, Zhang C. Effects of Pectus Excavatum on the Spine of Pectus Excavatum Patients with Scoliosis. J Healthc Eng. 2017;2017:5048625. doi: 10.1155/2017/5048625. Epub 2017 Jul 3. PMID 29065615
- [Result] Tomaszewski R, Wiktor L, Machala L. Evaluation of thoracic vertebrae rotation in patients with pectus excavatum. Acta Orthop Traumatol Turc. 2017 Jul;51(4):284-289. doi: 10.1016/j.aott.2017.03.005. Epub 2017 Jun 16. PMID 28624480
- [Result] Tauchi R, Kawakami N, Tsuji T, Ohara T, Suzuki Y, Saito T, Nohara A. Evaluation of thoracic factors after scoliosis surgery in patients with both scoliosis and pectus excavatum. Eur Spine J. 2018 Feb;27(2):381-387. doi: 10.1007/s00586-016-4753-4. Epub 2016 Aug 27. PMID 27568387
- [Result] Alaca N, Yuksel M. Comparison of physical functions and psychosocial conditions between adolescents with pectus excavatum, pectus carinatum and healthy controls. Pediatr Surg Int. 2021 Jun;37(6):765-775. doi: 10.1007/s00383-021-04857-7. Epub 2021 Jan 16. PMID 33454849
- [Result] Iscan M, Kilic B, Turna A, Kaynak MK. The effect of minimally invasive pectus excavatum repair on thoracic scoliosis. Eur J Cardiothorac Surg. 2020 Oct 30:ezaa328. doi: 10.1093/ejcts/ezaa328. Online ahead of print. PMID 33123728
- [Result] Tauchi R, Suzuki Y, Tsuji T, Ohara T, Saito T, Nohara A, Morishita K, Yamauchi I, Kawakami N. Clinical Characteristics and Thoracic factors in patients with Idiopathic and Syndromic Scoliosis Associated with Pectus Excavatum. Spine Surg Relat Res. 2018 Jan 27;2(1):37-41. doi: 10.22603/ssrr.2017-0027. eCollection 2018. PMID 31440644
- [Result] van Es LJM, van Royen BJ, Oomen MWN. Clinical significance of concomitant pectus deformity and adolescent idiopathic scoliosis: systematic review with best evidence synthesis. N Am Spine Soc J. 2022 Jun 25;11:100140. doi: 10.1016/j.xnsj.2022.100140. eCollection 2022 Sep. PMID 35814492
- [Result] Alaca N, Cagri Aslan D, Alaca I, Yuksel M. The psychometric properties of the Turkish version of the pectus carinatum body image quality of life questionnaire. Pediatr Surg Int. 2022 Jun;38(6):833-842. doi: 10.1007/s00383-022-05119-w. Epub 2022 Apr 7. PMID 35389073